CLINICAL TRIAL: NCT04482218
Title: Comparison Between the Old Diagnostic Tools for Paediatric Undernutrition and the New HAS 2019 Recommendations
Brief Title: Comparison Between the Old Diagnostic Tools for Paediatric Undernutrition and the HAS Recommendations
Acronym: EDEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0391
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Undernutrition
Keywords: Nutrition; Antromopemtric data; Pediatry
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Undernutrition is a widely under-diagnosed public health problem, including in pediatrics department. Undernutrition prevalence in pediatrics departments is about 15 to 20%.

Until now, there has been no national consensus on the criteria to be used to diagnose paediatric undernutrition. Until now, assessment focused on a range of non-consensus arguments that allowed the health care team to make its diagnosis. So, in the absence of well-defined criteria, diagnosis was based in part on experience and assesment team.

Since November 2019, the French High Authority of Health (Haute Authorité de Santé - HAS) has suggested recommendations to standardize pediatric undernutrition diagnosis.

The investigators offer to evaluate undernutrition prevalence differences diagnosed according to new HAS criteria compared to the previous diagnostic methodology.

The investigator's secondary aim is to identify profiles of children who do match between the two diagnostics methods.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort without change in care.

Following classic patient admission in involved departments, the investigating team moves to the department to collect data.

The measurements and informations collected are no different from those taken in the context of normal care.

All anthropometric measurements correspond to recommendations of good practice. Anthropometric measurements will be carried out by the healthcare team.

With collected data the investigators will evaluate undernutrition for each child, according to the 2 diagnostics methods.

For any diagnosis of undernutrition, the department dietician will be alerted so that the patient can be taken care of so it is done normally.

Data collected are as follows:

Simple demographic characteristics: Age, sex, departmentsand principal diagnosis Anthropometry: weight, height, brachial perimeter, head circumference Birth weight and date of term of pregnancy. Clinical history: all pathologies or clinical events that may be related to a weight variation.

Assessment of ingesta. A non-opposition will be asked

ELIGIBILITY:
Inclusion criteria:

* Patient under 18 years old (HAS 2019)
* Patient admitted to short and long-stay pediatric services at Montpellier University Hospital, other than maternity, neonatal, palliative care or resuscitation and rehabilitation department.

Exclusion criteria:

* Parental or child opposition
* Legal guardian unable to express consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 admitted for hospitalization in the pediatric deparment of the Montpellier University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison between HAS 2019 undernutrition criteria and previous diagnostic methodology | 2 month
  Comparison between HAS 2019 undernutrition criteria and previous diagnostic methodology

SECONDARY OUTCOMES:
Identified profiles of children who do match between the two diagnostics methods | 2 month
  Identified profiles of children who do match between the two diagnostics methods

CONTACTS AND LOCATIONS:
Overall Officials: Antoine AVIGNON, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC